CLINICAL TRIAL: NCT02034032
Title: A Randomized Controlled Trial of Regenexx™ SD Versus Exercise Therapy for Treatment of Knee Osteoarthritis With Historical Comparison to Total Knee Arthroplasty
Brief Title: Regenexx™ SD Versus Exercise Therapy for Treatment of Knee Osteoarthritis With Historical Comparison to TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MM-03-K
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Arthritis; TKA; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regenexx SD (Active Comparator): Regenexx-SD (Same Day) is a bone marrow based injection procedure.
  Interventions: Procedure: Regenexx SD
- Exercise Therapy (Active Comparator): Subjects in the Exercise Therapy group will attend an initial session with a trained Physical Therapist. During that session the physical therapist will instruct the subject in a home exercise program and instructions about activity limitations. The subject's progress will also be followed by the Physical Therapist during the 6 week follow-up visit with further instructions provided.
  Interventions: Behavioral: Exercise Therapy

INTERVENTIONS:
Procedure: Regenexx SD — stem cell treatment
  Arms: Regenexx SD
Behavioral: Exercise Therapy — exercise therapy control
  Arms: Exercise Therapy

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Regenexx SD compared to Exercise Therapy at three months. Historical comparison will be made to Total Knee Arthroplasty for treatment of knee osteoarthritis at 1 and 2 years.

DETAILED DESCRIPTION:
The study is single center, prospective, randomized, controlled trial to include 50 subjects, 25 treated with Regenexx SD and 25 treated with Exercise Therapy for treatment of knee osteoarthritis. Subjects will be enrolled within 60 days prior to Regenexx-SD injection or initiation of Exercise Therapy and take part in follow-up visits for two years following treatment. A preoperative visit will occur at the time of enrollment; follow-up visits will occur at the clinical site at 6 weeks, 3 months, 6 months, 12 months, and 24 months post injection.

Subjects in the control, exercise therapy arm, will have the opportunity to cross-over to the study treatment arm at or after the 3 month visit and then continue to be followed through 24 months.

Subjects will complete the study following the 2 year follow-up visit. They will be withdrawn from the study prematurely if a revision occurs.

The study subjects will be compared to a historical total knee arthroplasty group. Data of the TKA group subjects will be reviewed retrospectively after it is retrieved from the clinical database. The TKA group will consist of patients who underwent TKA for knee osteoarthritis. The inclusion criteria of age and BMI will be applied to these subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the IRB approved Informed Consent
2. Ages 18 to 70
3. Diagnosis of Knee osteoarthritis
4. Kellgren-Lawrence Grade 2 or 3 on X-Ray
5. BMI of <30
6. Minimum flexion to 110 degrees
7. Varus under 12 degrees/Valgus under 15 degrees
8. Instability in any plane less than 2 mm translation
9. ACL intact and no history of ACL reconstruction
10. Knee Society 100 point score > 65
11. If bilateral arthritis, subject must be able and willing to delay treatment of the second side for at least 6 months
12. Candidate is able to follow Regenexx medication guidelines
13. Patient agrees to return for periodic assessment protocol
14. Patient must execute all required documents
15. Patient must be appraised of Clinical Trial

Exclusion Criteria:

1. History of infection of the joint in the last five years
2. Intra-articular PRP, steroid or viscosupplementation in the last three months
3. Previous knee surgery within the last 6 months
4. Flexion contracture over 15 degrees
5. Low back pain with radiculopathy or with "significant" radiographic changes
6. History of immunosuppressive or chemotherapy in the last five years
7. Systemic neurological disease
8. HIV positive or chronic hepatitis
9. Any significant co-morbidity that in the opinion of the investigator should exclude the subject from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Knee Society Scores | 3 months
  Mean difference of Knee Society Scores for assessment and function between the treatment groups measured at 3 months

SECONDARY OUTCOMES:
KSS means difference between Regenexx SD and historical TKA data | 1 year
  The KSS means difference between Regenexx SD and historical TKA data measured at 1 year
KSS means difference between Regenexx SD and historical TKA data | 2 year
  The KSS means difference between Regenexx SD and historical TKA data measured at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Sheinkop, M.D., Principal Investigator — Regenerative Pain Center
Locations (1):
- Regenerative Pain Center; Weil Foot, Ankle and Orthopedic Institute, Des Plaines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Centeno C, Sheinkop M, Dodson E, Stemper I, Williams C, Hyzy M, Ichim T, Freeman M. A specific protocol of autologous bone marrow concentrate and platelet products versus exercise therapy for symptomatic knee osteoarthritis: a randomized controlled trial with 2 year follow-up. J Transl Med. 2018 Dec 13;16(1):355. doi: 10.1186/s12967-018-1736-8. PMID 30545387